CLINICAL TRIAL: NCT03830892
Title: Effects of E-Cigarette Power and Nicotine Content in Dual Users and Vapers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to COVID
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HM20012696; 2U54DA036105 (NIH)
Record Dates: First submitted 2019-01-14; First posted 2019-02-05 (Actual); Results first posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Electronic Cigarettes
MeSH Terms: conditions — Vaping | interventions — Nicotine; Tobacco Products

STUDY DESIGN:
Intervention Model Description: We will recruit two populations of e-cigarette users: exclusive e-cigarette users and dual users of e-cigarettes and tobacco cigarettes.
  All participants complete 5 within-subject laboratory conditions that each last 4 hours. Conditions (sessions) differ by the tobacco product used: 1) e-cigarette with low device power, low nicotine mg/ml; 2) e-cigarette with low device power, high nicotine mg/ml; 3) e-cigarette with high device power, low nicotine mg/ml; 4) e-cigarette with high device power, high nicotine mg/ml; and 5) own brand e-cigarette/cigarette.
  The first four sessions are latin-square-ordered and the last session for all participants will be their own brand cigarette/e-cigarette depending on the population. For dual users, we will counter-balance own brand condition product assignment (cigarette vs. e-cigarette). Conditions will differ in the presentation of primary outcomes (task order) which will be counterbalanced.
Who Masked: Participant
Masking Description: Participants will be blinded to their condition (power level and nicotine concentration) used in each session, except during their 'own brand' session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-cigarette User (Exclusive) (Active Comparator): Other: E-cigarette Lab Session 15 watts, 10 mg nicotine Other: E-cigarette Lab Session 15 watts, 30 mg nicotine Other: E-cigarette Lab Session 30 watts, 10 mg nicotine Other: E-cigarette Lab Session 30 watts, 30 mg nicotine Other: Own Brand Session - E-cigarette
  Interventions: Other: E-cigarette Lab Session 15 watts, 10 mg nicotine; Other: E-cigarette Lab Session 15 watts, 30 mg nicotine; Other: E-cigarette Lab Session 30 watts, 10 mg nicotine; Other: E-cigarette Lab Session 30 watts, 30 mg nicotine; Other: Own Brand Session - E-cigarette
- Dual User (Active Comparator): Other: E-cigarette Lab Session 15 watts, 10 mg nicotine Other: E-cigarette Lab Session 15 watts, 30 mg nicotine Other: E-cigarette Lab Session 30 watts, 10 mg nicotine Other: E-cigarette Lab Session 30 watts, 30 mg nicotine Other: Own Brand Session - E-cigarette/Cigarette
  Interventions: Other: E-cigarette Lab Session 15 watts, 10 mg nicotine; Other: E-cigarette Lab Session 15 watts, 30 mg nicotine; Other: E-cigarette Lab Session 30 watts, 10 mg nicotine; Other: E-cigarette Lab Session 30 watts, 30 mg nicotine; Other: Own Brand Session - E-cigarette; Other: Own Brand Session - E-cigarette/Cigarette

INTERVENTIONS:
Other: E-cigarette Lab Session 15 watts, 10 mg nicotine — E-cigarette paired with low nicotine, low device power
Other: E-cigarette Lab Session 15 watts, 30 mg nicotine — E-cigarette paired with low nicotine, low device power
Other: E-cigarette Lab Session 30 watts, 10 mg nicotine — E-cigarette paired with low nicotine, low device power
Other: E-cigarette Lab Session 30 watts, 30 mg nicotine — E-cigarette paired with low nicotine, low device power
Other: Own Brand Session - E-cigarette — E-cigarette paired with own brand liquid and preferred power
Other: Own Brand Session - E-cigarette/Cigarette — Own brand cigarette OR E-cigarette paired with own brand liquid and preferred power
  Arms: Dual User

SUMMARY:
This study aims to understand the effects of device power and nicotine concentration on the likelihood that someone would use or abuse e-cigarettes.

ELIGIBILITY:
Inclusion Criteria:

* healthy (determined by self-report)
* between the ages of 21-55
* willing to provide informed consent
* able to attend the lab and abstain from tobacco/nicotine as required and must agree to use designated products according to study protocol

Exclusion Criteria:

* Women if they are breast-feeding or test positive for pregnancy (by urinalysis) at screening.

Some study details about the eligibility criteria are purposely omitted at this time to preserve scientific integrity. Full details will be posted at the conclusion of the study.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Cobb (Amey), PhD, Principal Investigator — Virginia Commonwealth University; Andrew Barnes, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Center for the Study of Tobacco Products, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] White AM, Bono RS, Lester RC, Underwood M, Hoetger C, Lipato T, Bickel WK, Cobb CO, Barnes AJ. The electronic nicotine delivery system (ENDS) purchase task: Are results sensitive to price framing? Exp Clin Psychopharmacol. 2023 Oct;31(5):895-901. doi: 10.1037/pha0000631. Epub 2022 Dec 8. PMID 36480388
- [Derived] Hoetger C, Bono RS, White AM, Barnes AJ, Cobb CO. The interaction of nicotine concentration and device power on electronic nicotine delivery system (ENDS) abuse liability among exclusive ENDS users and dual users of ENDS and combustible cigarettes. Exp Clin Psychopharmacol. 2022 Dec;30(6):973-982. doi: 10.1037/pha0000523. Epub 2021 Oct 14. PMID 34647773

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each participant will participate in 6 sessions. Sessions differ by the tobacco product used (see study arms). The sessions are ordered by latin-square; however, session order was NOT expected to change any outcomes and order effects are not relevant to the study. Therefore all outcome data was merged and analyzed only by arm and session without regard to order.
Period: Overall Study
Arm/Group | E-cigarette User (Exclusive) | Dual User
Started | 25 | 23
15 Watts, 10 mg Nicotine | 19 | 17
15 Watts, 30 mg Nicotine | 19 | 17
30 Watts, 10 mg Nicotine | 19 | 17
30 Watts, 30 mg Nicotine | 19 | 17
Own Brand (Exclusive e-cigarette users only used e-cigarettes during own brand session, dual users used either their cigarettes and e-cigarettes. Completion of either one considered a milestone depending on study arm) | 19 | 17
Completed | 19 | 17
Not Completed | 6 | 6
Not completed — Physician Decision | 2 | 3
Not completed — Study terminated due to COVID | 4 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: Protocol was changed after study completion by 4 Dual Users so results are not being reported on those participants due to the protocol changes.
Groups:
- Total: Total of all reporting groups
Arm/Group | E-cigarette User (Exclusive) | Dual User | Total
Number analyzed (Participants) | 19 | 13 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.53 (7.53) | 29 (6.84) | 28.13 (7.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 13 | 7 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 18 | 12 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Middle Eastern | 0 | 1 | 1
  Black or African American | 3 | 3 | 6
  White | 13 | 8 | 21
  More than one race | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 19 | 13 | 32

OUTCOME MEASURES:

1. Primary Outcome: Breakpoint of Drug Purchase Tasks (DPT)
Description: The DPTs will yield measures of willingness to pay and measures of price sensitivity for session-specific tobacco products. Choices made during this task are not reinforced during the session. Each DPT will be completed once per study session (either 90 minutes or approximately 180 minutes into the session, timing varies based on task order presentation and potentially choices made in tasks presented prior to this task).
Time Frame: Up to 180 minutes
Population: Protocol was changed after study completion by 4 Dual Users so results are not being reported on those participants.
Measure: Mean (Standard Deviation); unit: US Dollars
Arm/Group | E-cigarette User (Exclusive) | Dual User
Number analyzed (Participants) | 19 | 13
US Dollars
  own brand e-cigarette | 3.95 (3.59) | 3.79 (3.09)
  30 watts, 30 mg/ml nicotine | 3.29 (3.73) | 4.43 (3.74)
  15 watts, 30 mg/ml nicotine | 3.51 (3.41) | 4.26 (3.63)
  30 watts, 10 mg/ml nicotine | 3.37 (3.43) | 4.23 (3.77)
  15 watts, 10 mg/ml nicotine | 3.74 (3.50) | 4.80 (3.86)

2. Primary Outcome: Breakpoint of Multiple Choice Procedure (MCP)
Description: The MCP will yield of measure of willingness to pay for session-specific tobacco products. One choice made during this task is reinforced (i.e., money or tobacco product is distributed). Completed once per study session (either 90 minutes or approximately 180 minutes into the session, timing varies based on task order presentation and potentially choices made in tasks presented prior to this task).
Time Frame: Up to 180 minutes.
Population: Protocol was changed after study completion by 4 Dual Users so results are not being reported on those participants.
Measure: Mean (Standard Deviation); unit: US Dollars
Arm/Group | E-cigarette User (Exclusive) | Dual User
Number analyzed (Participants) | 19 | 13
US Dollars
  Own brand e-cigarette | 3.05 (2.92) | 2.90 (2.99)
  30 watts, 30 mg/ml nicotine | 2.51 (3.18) | 2.36 (2.41)
  15 watts, 30 mg/ml nicotine | 2.56 (2.93) | 2.51 (1.98)
  30 watts, 10 mg/ml nicotine | 2.63 (2.98) | 2.10 (2.06)
  15 watts, 10 mg/ml nicotine | 2.35 (2.13) | 2.23 (2.34)

3. Primary Outcome: Effort for Product Puffs With the Progressive Ratio Task (PRT)
Description: The PRT will yield a measure of willingness to work for session-specific tobacco products (via number of times a space bar is pressed to earn puffs) by measuring the number of puffs self-administrated. Completed once per study session (either 90 minutes or approximately 180 minutes into the session, timing varies based on task order presentation and potentially choices made in tasks presented prior to this task).
Time Frame: Up to 180 minutes.
Population: Protocol was changed after study completion by 4 Dual Users so results are not being reported on those participants.
Measure: Mean (Standard Deviation); unit: e-cigarette puffs
Arm/Group | E-cigarette User (Exclusive) | Dual User
Number analyzed (Participants) | 19 | 13
e-cigarette puffs
  own brand e-cigarette | 4.95 (1.54) | 4.54 (1.56)
  30 watts, 30 mg/ml nicotine | 4.74 (1.88) | 4.54 (1.76)
  15 watts, 30 mg/ml nicotine | 4.58 (1.77) | 4.38 (2.06)
  30 watts, 10 mg/ml nicotine | 5.58 (1.68) | 5.38 (1.56)
  15 watts, 10 mg/ml nicotine | 4.89 (1.59) | 4.77 (1.92)

4. Other Pre Specified Outcome: Subjective Measures of Nicotine Abstinence Symptoms
Description: Measures of related to nicotine abstinence symptoms and nicotine side effects will be measured during each study session.
Time Frame: First measure given, regardless of task order, 90 minutes into each session
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Subjective Measures of Nicotine Abstinence Symptoms
Description: as for outcome 4
Time Frame: Third measure given during each session, approximately 120 minutes into each session (timing dependent on choices made in tasks presented prior to this measure).
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Subjective Measures of Nicotine Abstinence Symptoms
Description: as for outcome 4
Time Frame: Fifth measure given during each session, approximately 180 minutes into each session (timing dependent on choices made in tasks presented prior to this measure).
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Subjective Measures of Nicotine Abstinence Symptoms
Description: as for outcome 4
Time Frame: Last measure given during each session, approximately 240 minutes into each session (timing dependent on choices made in tasks presented prior to this measure).
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Heart Rate
Description: Heart rate (measured in bpm)
Time Frame: Recorded throughout each 4 hour study session using automated software every 10 seconds.
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Systolic Blood Pressure
Description: Blood pressure (measured in mm)
Time Frame: Recorded throughout each 4 hour study session using automated software every 5 minutes.
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in Diastolic Blood Pressure
Description: and blood pressure (measured in hg)
Time Frame: Recorded throughout each 4 hour study session using automated software every 5 minutes.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Data were collected during laboratory visits, approximately over 3 weeks; no follow up data collection occurred.
Description: Protocol was changed after study completion by 4 Dual Users so results are not being reported on those participants.
  All adverse events occurred in between study sessions (i.e., while participants were not receiving the intervention). Because effects of interventions end as soon as the intervention ends, adverse events occurring in between sessions are not related to the intervention and data about prior nor current session details was not stored with adverse events data.
Arm/Group | E-cigarette User (Exclusive) | Dual User
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/13
Other Adverse Events (participants affected / at risk) | 3/19 | 7/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E-cigarette User (Exclusive) (N=19) | Dual User (N=13)
Hospitalization (Surgical and medical procedures) | 1 (1) | 0 (0) — Unrelated hospitalization
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E-cigarette User (Exclusive) (N=19) | Dual User (N=13)
Worsening cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-06-16): https://cdn.clinicaltrials.gov/large-docs/92/NCT03830892/Prot_001.pdf
  • Statistical Analysis Plan (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT03830892/SAP_002.pdf
  • Informed Consent Form (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT03830892/ICF_000.pdf